CLINICAL TRIAL: NCT02751099
Title: Bone Metabolism and Cardiovascular Risk After Kidney Transplant in Adult Patients
Brief Title: Bone and Cardiovascular Disease After Kidney Transplant
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor
Other Study IDs: CHLC.CI363.2016
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Chronic Renal Insufficiency; Disorder Related to Renal Transplantation; Metabolic Bone Diseases; Vascular Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bone Diseases, Metabolic; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and bone biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- de novo renal transplanted patients: renal transplanted patients
  Interventions: Other: transplanted patients

INTERVENTIONS:
Other: transplanted patients — bone biopsy, echocardiogram, blood samples

SUMMARY:
Bone disorder is a significant problem in chronic kidney disease (CKD), becoming almost universal in stage 5 CKD patients. Besides the healthcare costs, bone disorder is associated with life-threatening complications, including fractures and cardiovascular (CV) events. Kidney transplantation provides circa 68% decrease in mortality and improves co-morbidity. Still, bone disease persists after transplantation.

The investigators hypothesize that bone-derived hormones can induce CV events in kidney transplanted patients. Therefore, early evaluation of the bone health is recommended, and prevention of its complications is required. Bone biopsy, an invasive and expensive method, is the gold standard for bone disorders diagnosis. Therefore, non-invasive predictors for bone disease are necessary. Classical biochemical markers of bone formation and resorption have shown a low sensitivity and low specificity. New markers, as fibroblast growth factor 23 (FGF23), and its cofactor klotho, and sclerostin are promising new markers for predicting CKD-associated bone and CV disease after transplantation.

This study assesses the phenotype of bone disease after transplantation (given by bone histology) and its correlation with serum FGF23, klotho and sclerostin, in order to evaluate its performance predicting CKD-associated bone and CV disease.

DETAILED DESCRIPTION:
BACKGROUND. Chronic kidney disease (CKD) affects millions of people worldwide. Cardiovascular (CV) events cause more than 50% of the mortality risk in CKD patients, and the relative excess mortality is observed in younger patients, below 45 years of age. Decreased renal function led to changes in biochemical parameters (calcium, phosphorus, PTH and vitamin D levels) and disturbed mineral metabolism, which translates into different bone disorders (related to bone turnover, mineralization, and volume) and all these are associated with extra-skeletal calcifications. Bone disease at any stage of CKD is associated with CV morbidity. This cross-talk between bone and vessels constitute a systemic syndrome known as CKD-mineral and bone disorder (CKD-MBD), that is thought to be one of the major non-traditional risk factors for the extremely high rate mortality observed in this disease.

CKD-MBD is classified into four major histological groups (in terms of turnover, mineralization and volume): hyperparathyroid bone disease (high turnover disease, with normal mineralization and variable volume); adynamic bone disease (low turnover disease, with normal mineralization and decreased bone volume); osteomalacia (low turnover disease, with reduced mineralization and with normal or high bone volume); and mixed renal osteodystrophy (reduced mineralization with or without increased bone formation).

Kidney transplantation is the treatment of choice for established stage 5 CKD. Even with correction of uremia, post-transplant MBD is frequent and reflects the pre-existing CKD-MBD, the effects of renal dysfunction after transplantation, and the effects and consequences of immunosuppression. Transplanted patients with CKD-MBD have reduced quality of life and require medical assistance for bone pain, fractures and CV events. Indeed, cardiovascular disease remains the leading cause of death after renal transplantation, still doubling risk of the general population.

The gold standard for the diagnosis of CKD-associated bone disease is bone biopsy, an expensive and invasive procedure. Non-invasive markers of bone disease presently lack sufficient specificity and sensitivity to allow the differential diagnosis of renal osteodystrophy. New biomarkers are needed and, osteocyte-derived factors, as FGF23 and sclerostin, are promising answers.

FGF23 acts as a phosphaturic hormone, a suppressor of vitamin D and has some non-consensual effect on parathyroid hormone (PTH). FGF23 has a specific receptor but needs a co-factor, klotho protein, to perform the majority of its functions. Serum klotho levels in CKD are low, influencing the resistance to FGF23 activity. What happens in transplanted patients is not yet totally understood; some studies pointed out for endothelial dysfunction and cardiovascular disease mediated by these factors in the transplant setting. Besides, graft loss and mortality were related with high serum levels of FGF23 and with bone mineral density loss but their relation with histological bone disease is unknown.

Sclerostin is a glycoprotein product of the SOST gene in osteocytes and acts as a negative regulator of bone metabolism. Various observations have shown that CKD patients have high sclerostin serum levels, thus its potential role in renal osteodystrophy. The correlation between serum levels of sclerostin and histomorphometric parameters of bone turnover, osteoblast number and function in renal transplanted patients is not yet known. The impact of high sclerostin levels on CV disease and mortality is yet to be determined.

Studies relating sclerostin levels with CV mortality in dialysis patients are inconsistent. Studies in renal transplanted patients are lacking.

AIMS. The investigators will study the relationship of the new osteocyte-derived biomarkers of bone disease, FGF23 (and klotho) and sclerostin, with bone histologic changes and CV events at baseline and one year after transplantation. If an association is to be found, the performance of the biomarkers as predictors of CKD-MBD will be determined. Non-contrast CT will allow us to validate Adragão score in a population of renal transplants, as this score is only validated for dialysis patients. We will study possible correlations between coronary artery calcification score and demographic characteristics of patients; laboratorial levels of FGF23, klotho, esclerostin, PTH, calcium, phosphorus, calcium x phosphorus, magnesium, LDL-colestherol, and albumin (both at T0 and T1), bone turnover, mineralization and volume (both at T0 and T1), and DXA results at 1 year. From these findings, we will try to discover potential new risk factors for vascular calcifications in renal transplant patients and potential pathophysiological mechanisms for this phenomenon.

METHODS. Prospective cohort study of a convenience, consecutive sample of de novo renal transplanted patients.

At recruitment, data will be collected on aetiology of CKD, presence of diabetes, hypertension, hyperparathyroidism, hepatitis virus, ovulation status for woman (menopause or not), active pre-transplant medication (with emphasis in vitamin D analogues, calcimimetics, and phosphate binders), echocardiography (M mode and 2D), Teresa Adragão score of vascular calcifications (hands and pelvis x-rays), HLA phenotype and mismatches, donor data (age, gender, cause of death), cold ischemia time.

Patients will be followed-up for 1 year, during which data will be recorded on immunosuppressive regimens (cumulative doses), CV events (myocardial infarction, congestive heart failure, arrhythmia), fractures, rejection episodes, graft loss (and its cause), and death (CV [fatal myocardial infarction, sudden death and fatal congestive heart failure], infection, malignancy or other). At the end of follow-up, echocardiogram (M mode and 2D) and scoring of vascular calcifications will be performed.

Serum creatinine, urea, ionogram, uric acid, calcium, phosphorus, magnesium, and bone alcaline phosphatase will be assessed using standard methods. PTH will be measured by immuno-chemiluminescence using a second-generation assay (Immulite 2000; Siemens Medical Solutions Diagnostics, Los Angels, CA). Vitamin D [25(OH)D and 1,25(OH)2D] will be measured with radioimmunoassay provided by IDS (Boldon, UK).

Two bone biopsies are proposed to each patient (just before the renal transplantation procedure, already on general anaesthesia, and circa 12 months after transplantation, with local anaesthesia). Bone biopsies will be made using a 7G trocar (Osteobell T), by manual puncture. After processing the bone fragment (fixation, dehydration and methylmethacrylate impregnation), routine staining will be used: von Kossa, Goldner trichrome, acid phosphatase (selective staining of osteoclasts), and Perls. Cortical bone will be evaluated separately from trabecular bone. Cortical bone volume and cortical thickness will be measured. Bone biopsies will be described for: bone remodelling and degree of cellular activation (specific score); efficacy of mineralization; quantification of possible metal deposits. In order to evaluate the rate of bone formation and rate of mineral deposition, the patient will be prescribed tetracycline hydrochloride, 500mg, 12/12 hours for three days, one month and one week before the 2nd bone biopsy or, in the case of live donor transplantation, before the 1st and 2nd bone biopsy.

At the same time point of the bone biopsies [at day 0 (pre-transplant) and nearly at month 12] serum levels of FGF23, and its cofactor Klotho, and sclerostin will be measured in the immunology lab of our hospital, according to the manufacturer's instructions. C-terminal FGF23 will be measured by sandwich ELISA (Immunotopics, San Clement, CA). Alfa-klotho will be measured by ELISA (IBL America, MN, USA). Sclerostin will be assessed by TECO Sclerostin EIA kit, which is a 96-well immune-capture ELISA (Sissach, Switzerland).

Comparisons between bone biopsies before and after transplantation will be assessed by paired t-test (if comparing scores) or by paired McNemar's test (after switching scores into categorical variables). Multivariable analysis adjusted for age, gender, diabetes, immunosuppressive regiments and/or its cumulative doses, and renal function will be performed to identify independent risk factors for the disease type and severity. In females, menopause will be considered as an effect modifier of bone volume.

Comparisons between FGF23, Klotho and sclerostin pre and post-transplant will be made by paired t-test, assuming normal distribution. Associations between FGF23, Klotho and sclerostin levels with demographic data and biochemical parameters in the two time-points will also be accessed with t-test, with Pearson test and linear regression, whenever applicable. A multivariable analysis will be executed to control for confounders (age, gender, diabetes, PTH, renal function, immunosuppressive regiments). Associations between FGF23, Klotho and sclerostin with bone turnover, mineralization and volume will be explored with regression models. The potential effects of FGF23 or sclerostin with CV health will be explored using regression models.

we are proposing to study as well vascular calcifications in post-transplant renal patients. For this, we will evaluate vascular calcifications by two different methods:

* Plain X-ray of the pelvis and hands for evaluation of vascular calcifications through Teresa Adragão score at day 0 and nearly at 12 months.
* Non-contrast CT in a low-radiation exposure technique, quantified using the Agatston method(26), performed nearly at 15 months after the renal transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for kidney transplantation.

Exclusion Criteria:

* mental retardation,
* liver-kidney transplantation.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: de novo renal transplanted patients, admitted to our renal transplantation unit.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Metabolic Bone Diseases | 12 months
  Histological pattern of bone disease
Cardiovascular disease | 12 months
  left ventricular hypertrophy, myocardial infarction, congestive heart failure, arrhythmia

SECONDARY OUTCOMES:
Bone fracture | 12 months
  Bone fracture
vascular calcification | 12 months
  hands and pelvis vascular calcification

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Carina Ferreira, MD, Principal Investigator — Nephrology Department, Centro Hospitalar de Lisboa Central
Locations (1):
- Nephrology Department, Centro Hospitalar de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferreira AC, Mendes M, Silva C, Cotovio P, Aires I, Navarro D, Caeiro F, Salvador R, Correia B, Cabral G, Nolasco F, Ferreira A. Biochemical Clusters as Substitutes of Bone Biopsies in Kidney Transplant Patients. Calcif Tissue Int. 2024 Mar;114(3):267-275. doi: 10.1007/s00223-023-01173-1. Epub 2024 Jan 22. PMID 38253933
- [Derived] Ferreira AC, Mendes M, Silva C, Cotovio P, Aires I, Navarro D, Caeiro F, Ramos R, Salvador R, Correia B, Cabral G, Nolasco F, Ferreira A. Improvement of Mineral and Bone Disorders After Renal Transplantation. Transplantation. 2022 May 1;106(5):e251-e261. doi: 10.1097/TP.0000000000004099. Epub 2022 Mar 8. PMID 35266925